CLINICAL TRIAL: NCT01492595
Title: Screening of Children in Household Contact With Adult TB Patients in Mbarara Hospital, Uganda: An Open Cohort of Children <5 Years in Contact With Newly Diagnosed Adult TB Cases in Mbarara Hospital
Brief Title: Screening of Children in Household Contact With Adult TB Patients in Mbarara Hospital, Uganda
Acronym: TBcontact
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Mbarara University of Science and Technology (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: Epicentre/MBA/2011/TBcontact
Record Dates: First submitted 2011-12-08; First posted 2011-12-15 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Tuberculosis
Keywords: contact
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed study aims to establish a pilot program through a prospective cohort study offering routine contact tracing, investigation and prophylaxis for LTBI, and treatment of TB disease to children <5 years living in the same household as adults diagnosed with smear/culture-positive pulmonary TB in Mbarara Regional Referral Hospital

DETAILED DESCRIPTION:
Because children with tuberculosis (TB) are usually smear-negative and therefore less infectious, they are generally not considered a public health risk. Up to 70% of children living in the same household with an adult with infectious TB will become infected, and more than 20% of them will develop active TB disease, usually within 12 months. The individual risk of developing disease once infected is highest in children <5 years. In addition, children under 5 years are at higher risk of developing disseminated forms of TB. The impact of childhood TB is worsened by co-infection with HIV. Contact tracing, investigation and prophylaxis of childhood contacts of adult TB cases are widely recommended but rarely practiced in developing countries. The World Health Organization recommends that all NTPs screen household contacts for symptoms of disease and offer isoniazid preventive therapy (i.e. daily isoniazid for at least 6 months) to children aged less than 5 years and to all HIV-infected children who are household contacts. In Mbarara, an area with a high incidence of TB, no program currently exists for the routine investigation of child contacts of adult pulmonary TB cases. Almost all child TB cases registered are found through the evaluation of symptomatic children, often long after the adult source-cases have been investigated and treated. The number of adult cases with pulmonary TB, together with the population structure in Mbarara (>50% of the total population being children) suggests that the number of childhood TB cases is probably higher than current hospital records indicate.

The proposed study aims to establish a pilot program through a prospective cohort study offering routine contact tracing, investigation and prophylaxis for LTBI, and treatment of TB disease to children <5 years living in the same household as adults diagnosed with smear/culture-positive pulmonary TB in Mbarara Regional Referral Hospital. The study will also generate much needed data on the utility of simple symptom-based screening of child contacts for TB disease in areas where access to radiological examination and tuberculin skin test are limited and on the efficacy and safety of IPT, in a region with a significant problem of HIV co-infection.

Children aged 1 month to 5 years living in the same household (a house or cluster of houses on the same plot) with a newly diagnosed adult case of smear and/or culture-positive TB will be eligible for the study. Children will undergo a physical examination, chest Xray, tuberculin skin test and specimen collection in case of symptoms. Children will then be classified as active TB, TB infected and non infected cases. TB infected and non infected children will receive 6 months isoniazid prophylaxis with monthly monitoring of acceptability and tolerability. A final clinical assessment will be performed at 9 months. A total of 577 children contacts will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Any child who has lived in the same household with the index case continuously for at least 2 weeks within the 3-month period immediately preceding the diagnosis of smear- positive or culture-positive TB in the index case.
* Informed consent signed by the parent or legal guardian
* Living within a 2-hour radius of Mbarara town

Exclusion Criteria:

* Child currently receiving anti-tuberculosis treatment
* Child has received a full course of anti-TB treatment within the last 6 months

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 month to 5 years living in the same household (a house or cluster of houses on the same plot) with a newly diagnosed adult case of smear and/or culture-positive TB will be eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of <5 year-old child contacts classified as active TB disease, LTBI or no infection | Baseline

SECONDARY OUTCOMES:
Number of children <5 years exposed to TB in the household of adult index cases | Baseline
Number of contacts identified as active TB basing on a symptom-based approach compared with those based on chest radiography | 9 months
Proportion of contacts with HIV co-infection classified as non infected, LTBI or active TB | 9 months
Median duration of exposure to symptomatic source case among the contacts in the various classes | Baseline
Association of various risk factors with the final classification of contacts after assessment | 9 months
Proportion of children with LTBI successfully treated (prevented from developing active TB disease) among HIV-infected and uninfected children | 9 months
Proportion of children with no TB infection or disease successfully treated (prevented from developing active TB disease or LTBI) | 9 months
Proportion of adverse events on treatment of TB disease, LTBI and TB exposure | 9 months
Adherence to IPT regimens | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Julius Kiwanuka, MD, Principal Investigator — Mbarara University of Science and Technology

IPD SHARING:
Plan to Share IPD: No